CLINICAL TRIAL: NCT05096975
Title: Comparative Study of the Personality Profile of Children and Adolescents With Attention Deficit Hyperactive Disorder (ADHD) With or Without Emotional Dysregulation
Brief Title: Personality Profile of Children and Adolescents With ADHD and With or Without Emotional Dysregulation
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0524
Record Dates: First submitted 2021-10-18; First posted 2021-10-27 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Attention Deficit Disorder; Emotional Dysfunction
Keywords: Personality traits; Children; Attention Deficit Hyperactivity Disorder; Emotion dysregulation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: ADHD without emotion dysregulation (Control group) The group is composed of children with ADHD and with a score ≤ 180 at the CBCL-A-A-A when combining the "Aggressive behaviors", "Anxiety/Depression" and "Attention" subscales.
  Interventions: Other: Evaluation of the CBCL-A-A-A and HiPIC in children with ADHD and with ED or without ED
- Deficit Emotion Self Regulation group: ADHD without moderate emotion dysregulation (Deficit Emotion Self Regulation group) The group is composed of children with ADHD and with a score ≥180 and ≤ 210 at the CBCL-A-A-A when combining the "Aggressive behaviors", "Anxiety/Depression" and "Attention" subscales.
  Interventions: Other: Evaluation of the CBCL-A-A-A and HiPIC in children with ADHD and with ED or without ED
- Dysregulation Profile Group: ADHD with severe emotion dysregulation (Dysregulation Profile Group) The group is composed of children with ADHD and with a score ≥ 210 at the CBCL-A-A-A when combining the "Aggressive behaviors", "Anxiety/Depression" and "Attention" subscales.
  Interventions: Other: Evaluation of the CBCL-A-A-A and HiPIC in children with ADHD and with ED or without ED

INTERVENTIONS:
Other: Evaluation of the CBCL-A-A-A and HiPIC in children with ADHD and with ED or without ED — The intervention involves the completion of two questionnaires by parents at child psychiatry unit of Montpellier University Hospital when children come to participate in a psychometric assessment or when parents or children participate in therapeutic group.
  All parents completed Child Behavior Checklist (CBCL; Achenbach & Rescorla, 2001), a 118-item questionnaire to measure emotional and behavior problems in 4 to 18-years-old children in the past six months and Hierarchical Personality Inventory for Children (HiPIC, Mervielde & De Fruyt, 1999, a 144-item questionnaire to obtain a profile of the personality of 6 to 12-year-old children.

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) is frequently associated with emotional dysregulation (ED). ED is characterized by excessive and inappropriate emotional reactions compared to social norms, uncontrolled and rapide shifts in emotion and attention focused on emotional stimuli.

According to research, there are strong correlations between personality traits and psychiatric disorder as ADHD. In a longitudinal study, the persistence of ADHD symptoms during adolescence is associated with high neuroticism, low agreeableness and low conscience. Studies show that these personality traits are factors of vulnerabilities for comordities associated with ADHD and are predictive of overall functioning difficulties. Studies show correlations between ADHD in childhood and personality disorders at adulthood .

ADHD is frequently associated with emotional dysregulation (ED) that is characterized by an inability to modulate emotional responses in a given context . ED is observed in 24% to 50% children with ADHD . Children with ADHD and ED are more likely to present a severe and complex symptomatology and are at risk for antisocial and bordeline personality disorders than children without ED. To date, there would be no studies which would have been interested in personality traits in children with ADHD and ED.

The main objective is to determine if children with ADHD and ED present from childhood traits of personality as low agreeableness, low conscience and high neuroticism that are predictive of personality disorders at adulthood. It would involve earl identification of children at increased risk of pejorative developmental trajectories.

The second objectives are:

* Improve understanding of the heterogeneity of ADHD symptom expression;
* Have a better understanding of the child's personalit and temperament traits to identify riks and protective factors;
* Identify children with ADHD with profiles at risk of personality disorders in order to adapt the care according to the child's needs.

ELIGIBILITY:
Inclusion criteria:

* Children and adolescents aged 7-12 years followed at Montpellier University Hospital ;
* Children and adolescents with a diagnostic of ADHD (diagnostics criteria from DSM-V);
* Children and adolescents benefiting from a multidisciplinary evaluation or therapeutic group at the child psychiatry unit of Montpellier University Hospital

Exclusion criteria:

- Family non-french speaking

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: * Children with a diagnostic of ADHD and followed at Montpellier University Hospital.
  * Children and adolescents aged between 7 and 12 years.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Rate of Score at the CBCL-A-A-A | 1 day
  Score at the CBCL-A-A-A when combining the "Aggressive behaviors", "Anxiety/Depression" and "Attention" subscales (Achenbach & Rescorla, 2001).
  Questionnaire measures emotional and behavior problem in 4 to 18 year-old children in the past months.

SECONDARY OUTCOMES:
Rate of Score of Hierachical Personality Inventory for Childen | 1 day
  Score of Hierachical Personality Inventory for Childen (HiPIC, Mervielde & De Fruyt, 1999), 144-item questionnaire to obtain a profile of the personality
  Questionnaire obtains a profile of personality of 6 to 12 year-old children.

CONTACTS AND LOCATIONS:
Overall Officials: Diane Purper-Ouakil, M.D., Ph. D., Study Director — UH Montpellier; Romo, PHD, Study Director — University Paris Nanterre
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC